CLINICAL TRIAL: NCT01186003
Title: Effectiveness of a Subcutaneously Administered Long-Acting Insulin Detemir Added to Insulin Drip Therapy as Compared With Standard Insulin Drip Treatment
Brief Title: Effectiveness of Adding Subcutaneous Long-Acting Detemir to Insulin Drip Therapy Compared With Standard Insulin Drip Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-0483
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Standard insulin drip therapy (No Intervention)
- Insulin drip and Detemir (Active Comparator): Detemir 0.25 units per kg body weight given subcutaneously every 24 hours while patients are receiving intravenous (IV) standard insulin drip therapy
  Interventions: Drug: Detemir

INTERVENTIONS:
Drug: Detemir — Detemir 0.25 units per kg body weight given subcutaneously every 24 hours while patients are receiving intravenous (IV) standard insulin drip therapy
  Other Names: Levimir
  Arms: Insulin drip and Detemir

SUMMARY:
The investigators anticipate that the use of Detemir will decrease the duration of an insulin drip, the dose of short-acting insulin in the drip, hospital and ICU (intensive care unit) length of stay, improve glycemic control, and prevent rebound hyperglycemias when the insulin drip is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic ketoacidosis (DKA) and hyperosmolar non-ketotic states, hyperglycemia with severe illness, pre-and postoperative states, nothing by mouth (NPO), as well as gastric (tube feeding) and parenteral nutritional requiring insulin drip.
* Patients with type 1 and type 2 diabetes mellitus (DM) will be included.
* Patient with both types of diabetes will be among those treated with insulin drip while being NPO, having severe concomitant illness or receiving enteral and parenteral nutrition
* Patients will be of age 19 to 80.

Exclusion Criteria:

* Inability to consent for the study for any reason including cognitive impairment secondary to hyperglycemia, presence of severe medical conditions requiring intubation, severe sepsis, hypothermia, and anticipated length of insulin drop 2 weeks and longer, pregnancy, Levemir allergy, and concurrent sulfonamide treatment

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Draznin, MD., Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Insulin Drip Therapy: Continuous IV insulin infusion without added detemir
Period: Overall Study
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.2) | 54.1 (16.2) | 53.26 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 11 | 12 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 12 | 13 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Rebound Hyperglycemia (Blood Glucose Levels Over 180 mg/dl)
Description: Number of participants exhibiting rebound hyperglycemia (blood glucose levels over 180 mg/dl)
Time Frame: within 48 hours of discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Number analyzed (Participants) | 14 | 16
Participants | 14 | 3

2. Secondary Outcome: Reduction in Duration of Insulin Drip Therapy and Reduction in Total and Average Per Hour Insulin Drip Dose
Time Frame: within one week of insulin drip therapy
Population: We have no information regarding whether this outcome measure was collected or analyzed. The PI has retired, and CU Clinical Research Administration has contacted the study team and PI on numerous occasions to try and obtain the data, but have not been able to do so. Therefore, this outcome measure cannot be reported.
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Reduction in ICU Length of Stay
Time Frame: within two weeks of hospitalization
Population: as for outcome 2
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Equal or Improved Diabetes Control
Time Frame: within two weeks of hospitalization
Population: as for outcome 2
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Reduction in Time to Get Back to Control of Glycemia (140-180 mg/dl) if Rebound Hyperglycemia Occurs
Time Frame: within one week post insulin drip
Population: as for outcome 2
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Week
Arm/Group | Standard Insulin Drip Therapy | Insulin Drip and Detemir
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

LIMITATIONS AND CAVEATS:
We have no information regarding whether many of the outcome measure were collected or analyzed. The PI has retired, and CU Clinical Research Administration has contacted the study team and PI on numerous occasions to try and obtain the data, but have not been able to do so. Therefore, several outcome measures cannot be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No